CLINICAL TRIAL: NCT06133075
Title: Using Mirabegron to Increase Blood Pressure in Patients With Postural Orthostatic Tachycardia Syndrome
Brief Title: Using Mirabegron to Increase BP in Patients With POTS
Acronym: RAISE BP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Peng-Sheng Chen, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002281
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; Chronic Orthostatic Intolerance; Syncope
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Syncope | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: All patients will receive mirabegron 50 mg or 25 mg orally for 8 weeks to determine their effects on blood pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 mg group (Active Comparator): Ten patients will receive 50 mg mirabegron for 8 weeks.
  Interventions: Drug: Mirabegron 50 MG
- 25 mg group (Active Comparator): Ten patients will receive 25 mg mirabegron for 8 weeks.
  Interventions: Drug: Mirabegron 25 MG

INTERVENTIONS:
Drug: Mirabegron 50 MG — 10 patients will receive drug for 8 weeks
  Other Names: Myrbetriq
  Arms: 50 mg group
Drug: Mirabegron 25 MG — 10 patients will receive drug for 8 weeks
  Other Names: Myrbetriq
  Arms: 25 mg group

SUMMARY:
This is a pilot dose-finding study to test the hypothesis that mirabegron increases systolic blood pressure (BP), prevents syncope/presyncope, and improves the quality of life (QOL), functional capacity, chest pain, and overactive bladder (OAB) symptoms in patients with postural orthostatic tachycardia syndrome (POTS) who have a documented history of hypotension inadequately responsive to conventional treatments. The American Heart Association funds this study.

DETAILED DESCRIPTION:
This is a pilot dose-finding study to test the hypothesis that mirabegron increases systolic blood pressure (BP), prevents syncope/presyncope, and improves the quality of life (QOL), functional capacity, chest pain, and overactive bladder (OAB) symptoms in patients with postural orthostatic tachycardia syndrome (POTS) who have a documented history of hypotension inadequately responsive to conventional treatments. The investigators will perform 24-hour ambulatory blood pressure monitoring (ABPM) and ambulatory skin sympathetic nerve activity (SKNA) recording using a Bittium Faros electrocardiogram (ECG) monitor, assess the number of syncope and presyncope episodes and determine the symptoms using validated questionnaires at baseline. The patients will then be given mirabegron (either 25 mg once daily or 50 mg once daily) for eight weeks. Afterward, the patient will return to the clinic for clinical assessments, complete questionnaires, ABPM, and ambulatory SKNA recording while still on treatment. Mirabegron will be stopped when the data collection is complete. Because mirabegron has a long half-life, the investigators will schedule a video visit with the patient 12 weeks after beginning the treatment and inquire about the patient's symptoms. The investigators will repeat all pertinent questionnaires at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Age > 18 years old.
3. Documented history of chronic (> 3 months) of orthostatic intolerance.
4. Diagnosis of syncope or pre-syncope and documented intermittent hypotension unresponsive to conventional life-style modification therapy.

   1. A history of syncope (complete loss of consciousness) or presyncope (the sensation that one is about to pass out).
   2. At least one documented hypotensive episode with systolic BP < 90 mmHg on 24-hr ABPM.
   3. Inadequate response to conventional therapies.

Exclusion Criteria:

1. Patients with other potential etiologies of syncope

   1. Sustained tachyarrhythmias other than sinus tachycardia. Specifically, patients with a diagnosis of atrial fibrillation, sustained (> 30 seconds) arrhythmias including paroxysmal supraventricular tachycardia, atrial flutter, ventricular tachycardia, ventricular fibrillation.
   2. Symptomatic bradycardia before pacemaker implantation.
2. Heart failure with either preserved or reduced ejection fraction.
3. Wolff Parkinson-White Syndrome.
4. Stroke within the past 6 months.
5. Any history of myocardial infarction.
6. Active thyrotoxicosis.
7. Any experimental medication concomitantly or within 4 weeks of participation in the study.
8. Patients < 18 years old because mirabegron is not approved by FDA for use in children.
9. People with a history of allergy to ECG electrodes or adhesive tape.
10. Patients with known contraindications or precautions to mirabegron.

    1. Hypertension
    2. Severe renal impairment (calculated CrCl < 30ml/min)
    3. Hepatic disease (Child-Pugh Class B)
    4. Pregnant or lactation
    5. Geriatric patients in long term care facilities
    6. Patients who are known to be allergic to mirabegron
    7. Patients taking drugs that are CYP2D6 substrates, such as midodrine. An extensive list can be found at the following website: https://drug-interactions.medicine.iu.edu/MainTable.aspx
11. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8 weeks
  Mirabegron changes the average systolic BP in 24-hr ABPM recording

SECONDARY OUTCOMES:
Syncope | 8 weeks
  Change of frequencies of syncope and presyncope
Hypotensive episode | 8 weeks
  Change of the hypotensive (systolic BP < 90 mmHg) episodes during wake time using ABPM
Duke Activity Status Index Questionnaire | 8 weeks
  Change of functional capacity score as measured by the Duke Activity Status index questionnaire
EQ-5D-5L Questionnaire | 8 weeks
  Change of health related QOL score using a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Seattle Angina Questionnaire (SAQ) | 8 weeks
  Change of QOL and symptoms of angina as measured by the SAQ based on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale.
Overactive Bladder symptoms | 8 weeks
  Change in OAB symptoms as measured by the OAB-q SF

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No